CLINICAL TRIAL: NCT01075451
Title: Antimicrobial Drug Use and Resistant Staphylococcus Aureus in a Network of Academic Medical Center Hospitals.
Brief Title: Antimicrobial Drug Use and Resistant Staphylococcus Aureus
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: University HealthSystem Consortium (Other); Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Other Study IDs: PT104711
Record Dates: First submitted 2010-02-23; First posted 2010-02-25 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Staphylococcus Aureus
Keywords: Staphylococcus aureus; Antimicrobial Stewardship; Antibacterial resistance; Vancomycin
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this investigation is to study the relationships between antimicrobial stewardship program efforts, antimicrobial drug use, and infection control efforts to the incidence rates of hospital acquired infections with Staphylococcus aureus in a sample of US academic medical center hospitals.

DETAILED DESCRIPTION:
Hospitalized patients can become infected with a variety of microorganisms, but infections caused by Staphylococcus aureus (i.e., "staph" infections) are particularly common. The main strategy to reduce the number of patients infected with Staph. aureus is to decrease cross-transmission from one patient to another. In addition, increasing evidence suggests that improvements in antimicrobial drug use--promoted by hospital Antimicrobial Stewardship programs (ASPs) -- may also favorably impact rates of Staph. aureus infections. While many Staphylococcal strains remain susceptible to an old drug called methicillin (methicillin-susceptible Staph aureus, or MSSA), many Staph. aureus are methicillin-resistant (MRSA). The drug of choice for MRSA has historically been vancomycin, and vancomycin is now the most commonly prescribed antibiotic in US teaching hospitals. Vancomycin-resistant Staph. aureus (VRSA) is still uncommon, but some Staph. aureus are developing "low level" resistance to vancomycin. These strains are often called S. aureus with MIC "creep" to vancomycin (SA-MICcreep), and Staphylococcus aureus with Heterogeneous Resistance to Vancomycin (hVISA), but the epidemiology, clinical significance and risk factors for these organisms are not well described. We will survey UHC participating hospitals to learn more about these organisms, the drug and ASP related risk factors, and whether hospitals are trying to identify these organisms.

ELIGIBILITY:
Inclusion Criteria:

* NA

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aggregate antibacterial drug use from adult inpatients at 60 UHC hospitals for 2006 - 2009
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2010-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Association between Antimicrobial Stewardship Program and Infection Control efforts, antibacterial drug use and rates of hVISA and other resistant staphylococci. | 2008 and 2009
  Rates of hVISA and Staph.aureus with MIC creep to vancomycin

CONTACTS AND LOCATIONS:
Overall Officials: Ron E Polk, Pharm.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University School ofPharamcy, Richmond, Virginia, United States

REFERENCES:
- [Background] Pakyz AL, Oinonen M, Polk RE. Relationship of carbapenem restriction in 22 university teaching hospitals to carbapenem use and carbapenem-resistant Pseudomonas aeruginosa. Antimicrob Agents Chemother. 2009 May;53(5):1983-6. doi: 10.1128/AAC.01535-08. Epub 2009 Mar 9. PMID 19273670
- [Background] Pakyz AL, MacDougall C, Oinonen M, Polk RE. Trends in antibacterial use in US academic health centers: 2002 to 2006. Arch Intern Med. 2008 Nov 10;168(20):2254-60. doi: 10.1001/archinte.168.20.2254. PMID 19001203
- [Background] Pakyz A, Powell JP, Harpe SE, Johnson C, Edmond M, Polk RE. Diversity of antimicrobial use and resistance in 42 hospitals in the United States. Pharmacotherapy. 2008 Jul;28(7):906-12. doi: 10.1592/phco.28.7.906. PMID 18576905
- [Background] MacDougall C, Polk RE. Variability in rates of use of antibacterials among 130 US hospitals and risk-adjustment models for interhospital comparison. Infect Control Hosp Epidemiol. 2008 Mar;29(3):203-11. doi: 10.1086/528810. PMID 18257689